CLINICAL TRIAL: NCT04555096
Title: A Pilot, Randomized, Placebo-Controlled Trial of GC4419 (Avasopasem Manganese) in Patients With Critical Illness Due to SARS-CoV-2 Infection (COVID-19)
Brief Title: A Trial of GC4419 in Patients With Critical Illness Due to COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants are no longer receiving intervention
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COV-4419-201
Record Dates: First submitted 2020-09-16; First posted 2020-09-18 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: COVID19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — avasopasem manganese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active GC4419 (Experimental): Arm A
  Interventions: Drug: GC4419
- Placebo (Placebo Comparator): Arm B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GC4419 — 180 Minute IV Infusion
  Other Names: Avasopasem
  Arms: Active GC4419
Drug: Placebo — 180 Minute IV Infusion
  Arms: Placebo

SUMMARY:
A Trial of GC4419 in Patients with Critical Illness due to COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age.
2. Ability to understand and the willingness to sign a written informed consent.
3. Laboratory-confirmed SARS-CoV-2 infection as determined by a positive PCR test documented prior to randomization
4. Requirement for intensive inpatient hospital care
5. Acute hypoxemic respiratory failure typifying ARDS
6. Adequate liver function
7. Use of effective contraception

Exclusion Criteria:

1. Expected survival for less than 48 hours after randomization
2. Child-Pugh stage C hepatic impairment and/or portal hypertension secondary to cirrhosis
3. Stage IV chronic kidney disease or end-stage kidney disease on maintenance hemodialysis
4. Requirement for extra-corporeal membrane oxygenation (ECMO)
5. Acute Myocardial Infarction (AMI)
6. Active bleeding requiring transfusion
7. Concurrent participation in another clinical trial of experimental treatment for SARSCoV-2
8. Female patients who are pregnant or breastfeeding
9. Requirement for concurrent treatment with nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Holmlund, MD, Study Chair — Study Chair
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Saint Louis University, St Louis, Missouri
  - Mercy Research, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson JOG, Jynge P, Ignarro LJ. May Mangafodipir or Other SOD Mimetics Contribute to Better Care in COVID-19 Patients? Antioxidants (Basel). 2020 Oct 10;9(10):971. doi: 10.3390/antiox9100971. PMID 33050459

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active GC4419 | Placebo
Started | 9 | 7
Completed | 4 | 2
Not Completed | 5 | 5
Not completed — Death | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the same.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active GC4419 | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.89) | 64.0 (11.28) | 63.3 (61.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: 28 Day All-cause Mortality
Description: Death rate of patients with critical illness due to COVID-19 28 days after initiation of therapy.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active GC4419 | Placebo
Number analyzed (Participants) | 9 | 7
Participants
  Alive | 5 | 3
  Death | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events collected from the baseline visit until 30 days after the last dose of GC4419/Placebo
Arm/Group | Active GC4419 | Placebo
All-Cause Mortality (participants affected / at risk) | 4/9 | 4/7
Serious Adverse Events (participants affected / at risk) | 5/9 | 4/7
Other Adverse Events (participants affected / at risk) | 8/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active GC4419 (N=9) | Placebo (N=7)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active GC4419 (N=9) | Placebo (N=7)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Propofol infusion syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Electrocardiogram QR prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin injury (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (General disorders) | 5 (5) | 1 (1)
Shock (General disorders) | 0 (0) | 1 (1)
Increase respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to the inability to enroll critically ill COVID 19 patients as the height of the pandemic was over and the sites that were open for enrollment to the clinical study were no longer treating these types of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04555096/Prot_SAP_000.pdf